CLINICAL TRIAL: NCT01985191
Title: A Phase 1 Study of Combination Therapy With SAR405838 and Pimasertib in Patients With Advanced Cancer
Brief Title: A Safety and Efficacy Study of SAR405838 and Pimasertib in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD13388; 2013-002325-33; U1111-1144-8349 (Other: UTN)
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — SAR405838; N-(2,3-dihydroxypropyl)-1-((2-fluoro-4-iodophenyl)amino)isonicotinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): SAR405838 and pimasertib in escalating doses
  Interventions: Drug: SAR405838; Drug: Pimasertib

INTERVENTIONS:
Drug: SAR405838 — Pharmaceutical form:capsule
  Route of administration: oral
Drug: Pimasertib — Pharmaceutical form: capsule
  Route of administration: oral

SUMMARY:
Primary Objectives:

To determine the recommended Phase 2 dose of SAR405838 / pimasertib combination therapy in patients with solid tumors.

To assess the anti-tumor activities of SAR405838 / pimasertib in patients with solid tumors.

Secondary Objectives:

To characterize the pharmacokinetic profile of SAR405838 and pimasertib.

To evaluate the pharmacodynamic effect of the SAR405838 and pimasertib.

To characterize genetic status in tumor tissue and circulating tumor DNA.

DETAILED DESCRIPTION:
The duration of the study for an individual patient will include a period to assess eligibility of up to 4 weeks, a treatment period of at least 6 weeks of study treatment, and an end-of-study visit at least 30 days (or until the patient receives another anti-cancer therapy, whichever is shorter) following the last administration of study drug.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of a solid tumor.
* Presence of locally advanced or metastatic disease with at least one measurable lesion.
* Ability to provide written informed consent. Evidence of a personally signed informed consent.

Exclusion criteria:

* Age <18 years.
* Eastern Cooperative Oncology Group performance status of >1.
* Inadequate functions of bone marrow, liver, and kidney.
* Positive pregnancy test in women of child-bearing potential.
* Pregnancy or breast-feeding.
* Extensive prior radiotherapy.
* The patient has retinal degenerative disease, history of uveitis, or history of retinal vein occlusion, or history of retinal detachment, or has medically relevant abnormalities identified on screening ophthalmologic examination.
* Prior history of myositis or rhabdomyolysis.
* Recent major surgery or trauma, unhealing/open wounds.
* The patient has had congestive heart failure, unstable angina, a myocardial infarction, cardiac conduction abnormality or pacemaker or a stroke within 3 months of entering the study.
* The patient has a baseline corrected QT interval (QTc) >480 ms or left ventricular ejection fraction (LVEF) <50% or less than the lower limit of normal.
* The patient has a previously-identified allergy or hypersensitivity to components of the study treatment formulations.
* Unwillingness or inability to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.
* Unwillingness, if not postmenopausal or surgically sterile, to abstain from sexual intercourse or employ an effective barrier or medical method of contraception during the study drug administration and follow-up periods.
* Recent history of acute pancreatitis.
* Clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that could affect the safety of the patient; alter the absorption of the study drugs; or impair the assessment of study results.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
SAR405838 (pimasertib) RP2D assessed by dose-limiting toxicities and pharmacological activities | 6 weeks for each patient at each dose level
Changes of tumor dimension by imaging | At least 3 months for each patient

SECONDARY OUTCOMES:
Overall safety profile of SAR405838 (pimasertib), number of participants with adverse events | Throughout the study
Pharmacokinetic parameters for both SAR405838 (pimasertib): the maximum concentration in blood (Cmax) | 3 months for each patient
Pharmacokinetic parameters for both SAR405838 (pimasertib): time to the maximum concentration (Tmax) | 3 months for each patient
Pharmacokinetic parameters for both SAR405838 (pimasertib): area under the curve (AUC), etc. | 3 months for each patient
Biomarker changes in response to SAR405838 (pimasertib) treatment | 3 months for each patient
Genetic status in tumor tissue | Baseline
Change of the genetic status of circulating tumor DNA | Baseline and until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- Investigational Site Number 250001, Villejuif, France
- Netherlands (3):
  - Investigational Site Number 528001, Amsterdam
  - Investigational Site Number 528003, Rotterdam
  - Investigational Site Number 528002, Utrecht

REFERENCES:
- [Derived] de Weger VA, de Jonge M, Langenberg MHG, Schellens JHM, Lolkema M, Varga A, Demers B, Thomas K, Hsu K, Tuffal G, Goodstal S, Mace S, Deutsch E. A phase I study of the HDM2 antagonist SAR405838 combined with the MEK inhibitor pimasertib in patients with advanced solid tumours. Br J Cancer. 2019 Feb;120(3):286-293. doi: 10.1038/s41416-018-0355-8. Epub 2018 Dec 26. PMID 30585255